CLINICAL TRIAL: NCT04844983
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Intralesional Injection of STP705 in Adult Patients With Cutaneous Squamous Cell Carcinoma in Situ (isSCC)
Brief Title: A Study to Evaluate Safety, Efficacy of Intralesional Injection of STP705 in Patients With isSCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sirnaomics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SRN-705-008
Record Dates: First submitted 2021-04-09; First posted 2021-04-14 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Squamous Cell Carcinoma in Situ
MeSH Terms: conditions — Squamous Intraepithelial Lesions | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Part 1: 40 subjects randomized in a 1:1:1:1 ratio to receive 6 weeks of treatment of placebo, 30 ug, 60 ug, or 90 ug of STP705. Enrollment will be temporarily stopped after the 40th subject. Interim Analysis will be done for dose response assessment and selection of the 2 doses for Part 2 of the study.
  Part 2: 60 additional subjects will be randomized in a 1:1:1 ratio to receive placebo or one of the 2 selected STP705 doses.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study. All subjects, investigators, and site staff (except unblinded pharmacist or designated site staff) in the study will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1: Arm A (Experimental): STP705 30 μg dose, intralesional injection, given once a week for 6 weeks.
  Interventions: Drug: STP705
- Part 1: Arm B (Experimental): STP705 60 μg dose, intralesional injection, given once a week for 6 weeks.
  Interventions: Drug: STP705
- Part 1: Arm C (Experimental): STP705 90 μg dose, intralesional injection, given once a week for 6 weeks.
  Interventions: Drug: STP705
- Part 1: Arm D (Other): Placebo (normal saline), intralesional injection, given once a week for 6 weeks.
  Interventions: Other: Placebo Saline
- Part 2: Arm A, B or C (Experimental): STP705 selected dose 1, intralesional injection, given once a week for 6 weeks.
  Interventions: Drug: STP705
- Part 2: Arm A or B or C (Experimental): STP705 selected dose 2, intralesional injection, given once a week for 6 weeks.
  Interventions: Drug: STP705
- Part 2: Arm D (Other): Placebo (normal saline), intralesional injection, given once a week for 6 weeks.
  Interventions: Other: Placebo Saline

INTERVENTIONS:
Drug: STP705 — The STP705 drug substance is composed of two siRNA oligonucleotides, targeting TGF-β1 and COX-2 mRNA respectively.
  Other Names: STP705 Powder for Injection
  Arms: Part 1: Arm A; Part 1: Arm B; Part 1: Arm C; Part 2: Arm A or B or C; Part 2: Arm A, B or C
Other: Placebo Saline — Normal Saline
  Arms: Part 1: Arm D; Part 2: Arm D

SUMMARY:
The purpose of this trial is to evaluate safety, tolerability and efficacy of various doses of STP705 administered as intralesional injection in subjects with cutaneous squamous cell carcinoma (in situ) skin cancer (isSCC).

DETAILED DESCRIPTION:
This is a two-part, double-blind, randomized, placebo-controlled study designed to evaluate safety and efficacy of various doses of STP705 administered as an intralesional injection in subjects with isSCC.

A total of up to 100 eligible subjects will be enrolled. Enrolled subjects will be randomly allocated to receive STP705 or placebo injection once weekly for 6 weeks.

After 6 weeks, the lesion will be excised.

In part 1 (dose ranging study): 40 subjects will be randomized to receive 1 of the 3 STP705 doses or placebo.

An interim analysis will be done after all subjects have completed end of treatment (EOT) visits to determine 2 selected dose levels of STP705 to be used in part of the study.

In part 2: 60 additional subjects will be randomized to receive 1 of the 2 selected doses (from part 1) or placebo.

In both parts at the End of Treatment (EOT), the lesion will be excised.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult ≥ 18 years of age.
2. Primary, histologically confirmed trunk or extremity (non- anogenital/-facial/-scalp) isSCC lesion suitable for excision with a minimum diameter of 0.5 cm and with a maximum diameter of 2.0 cm.
3. Histological diagnosis made no more than 6 months prior to the screening visit.
4. No other dermatological disease in the isSCC target site or surrounding area, which in the opinion of the investigator, could interfere with the study.
5. Willing to refrain from using non-approved lotions or creams on the target site and surrounding area during the treatment period.
6. Willing to refrain from exposure to excessive direct sunlight or ultraviolet light and to avoid the use of tanning parlors for the duration of the study.
7. Laboratory values for the tests (listed in the Study Schedule) within the reference ranges as defined by the central laboratory, or "out of range" test results that are clinically acceptable to the investigator.
8. Ability to follow study instructions and likely to complete all study requirements.
9. Written informed consent obtained, including consent for tissue to be examined and stored by the Central Histology Lab.
10. Written consent to allow photographs of the target isSCC lesion to be used as part of the study data and documentation.
11. For females of childbearing potential, a negative pregnancy test at screening and using an acceptable form of birth control (oral / implant/ injectable/ transdermal contraceptives, intrauterine device, condom, diaphragm, abstinence, or a monogamous relationship with a partner who has had a vasectomy).

Exclusion Criteria:

1. Pregnant, lactating, or planning to become pregnant.
2. Presence of known or suspected systemic cancer.
3. Histological evidence of severe squamous metaplasia, infiltrative, desmoplastic or micronodular growth patterns in the biopsy specimen.
4. History of recurrence of the target isSCC lesion.
5. Concurrent disease or treatment that suppresses the immune system.
6. Patients with baseline QTC > 480 msec using Frederica's formula.
7. Chronic medical condition that in the judgment of the investigator(s) would interfere with the performance of the study or would place the patient at undue risk.
8. Known sensitivity to any of the ingredients in the study medication including an allergy to trehalose.
9. Use of a tanning bed or other excessive or prolonged exposure to ultraviolet light or direct sunlight during the study.
10. Treatment with systemic chemotherapeutic agents within the 6 months prior to the screening visit.
11. Use of systemic retinoids within the 6 months prior to the screening period.
12. Treatment with systemic immunomodulators or immunosuppressants within the 6 months prior to the screening period.
13. Use of topical immunomodulators within 2 cm of the target isSCC lesion within the 4 weeks prior to the screening period.
14. Treatment with the following topical agents within 2 cm of the target isSCC lesion within the 4 weeks prior to the screening visit: aminolevulinic acid, 5-fluorouracil, corticosteroids, retinoids, diclofenac, ingenol mebutate, or imiquimod.
15. Treatment with liquid nitrogen, surgical excision or curettage within 2 cm of the target isSCC lesion during the 4 weeks prior to the screening visit.
16. Evidence of current chronic alcohol or drug abuse.
17. Current enrollment in an investigational drug or device study or participation in such a study within 4 weeks of the screening visit.
18. In the investigator's opinion, evidence of unwillingness, or inability to follow the restrictions and requirements of the protocol and complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with histological clearance of treated isSCC lesion | 6 weeks
  Proportion of participants with histological clearance of treated isSCC lesion at the End of Treatment (EOT).

SECONDARY OUTCOMES:
Change in size of the treated isSCC lesion | 6 weeks
  Change in size of the treated isSCC lesion over the 6-week treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nestor, MD, Principal Investigator — Center for Clinical and Cosmetic Research; David Goldberg, Principal Investigator — Schweiger Dermatology Group; Michael Gold, MD, Principal Investigator — Tennessee Clinical Research; Edward Lain, MD, Principal Investigator — Austin Institute for Clinical Research; Kenneth Beer, MD, Principal Investigator — Research Institute of the Southeast LLC; Brenda LaTowsky, MD, Principal Investigator — Investigate MD; Edward Primka, MD, Principal Investigator — Dermatology Associates of Knoxville; Girish Munavalli, MD, Principal Investigator — Dermatology, Laser and Vein Specialists of the Carolinas; Brian Jiang, MD, Principal Investigator — University of California, San Diego; Megan Couvillion, MD, Principal Investigator — SBA Dermatology; Mark Ling, MD, Principal Investigator — Medaphase Inc
Locations (7):
- United States (7):
  - Investigate MD, Scottsdale, Arizona
  - Center for Clinical and Cosmetic Research, Aventura, Florida
  - Research Institute of the Southeast LLC, West Palm Beach, Florida
  - Dermatology, Laser and Vein Specialists of the Carolinas, Charlotte, North Carolina
  - Dermatology Associates of Knoxville, Knoxville, Tennessee
  - Tennessee Clinical Research, Nashville, Tennessee
  - Austin Institute for Clinical Research, Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: No